CLINICAL TRIAL: NCT07325747
Title: Immediate Versus Delayed Surgical Reconstruction of Peri-implantitis Intra-bony Defects: A Parallel-arm, Assessor-blind, Randomized, Controlled Clinical Trial
Brief Title: Immediate Versus Delayed Surgical Reconstruction of Peri-implantitis Intra-bony Defects.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Purnima S. Kumar, Professor and Chair of the Department of Periodontics and Oral Medicine, School of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00235330; AWD029397 (Other Grant/Funding Number: osteology Foundation)
Record Dates: First submitted 2025-12-10; First posted 2026-01-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Peri Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Regeneration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The subjects will receive treatment consisting of surgical defect debridement and decontamination, followed by intra-bony defect reconstruction via immediate guided bone regeneration (GBR).
  Interventions: Procedure: Simultaneous peri-implant debridement and regeneration
- Test Group (Experimental): The subjects will receive a two-stage treatment consisting of the surgical removal of peri-implant granulation tissue and pocket epithelium. After 4-6 weeks, they will undergo surgical defect debridement and decontamination, followed by intra-bony defect reconstruction via immediate guided bone regeneration (GBR).
  Interventions: Procedure: Staged peri-implant debridement and regeneration

INTERVENTIONS:
Procedure: Staged peri-implant debridement and regeneration — Peri-implant debridement will be carried our in visit one and will be followed by a second surgery for regeneration
  Arms: Test Group
Procedure: Simultaneous peri-implant debridement and regeneration — The peri-implant defect will be debrided and regenerated at the same visit.
  Arms: Control Group

SUMMARY:
The purpose of this study is to test the comparative efficacy of two surgical approaches (immediate versus delayed GBR) for the surgical reconstruction of peri-implantitis intra-bony defects in terms of the clinical, radiographical, histological, volumetric, microbiological, and patient-reported outcomes.

The investigators hypothesize that in certain clinical situations, treatment of peri-implantitis intra-bony defects with the use of a compound bone grafting material (mixture of allogenic bone substitutes) and a non-resorbable barrier membrane and following a delayed approach (test group) with initial phase of defect decontamination and initial healing phase would yield superior outcomes to that of the conventional approach (control group) of defect decontamination and regeneration at the same clinical visit while also significantly enhancing patient-reported outcomes:

H0: There is no difference between the two mentioned approaches in terms of the treatment outcomes. H1: There is a significant difference, favoring the delayed approach compared to the immediate reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adults
* Age ≥ 18 years
* The patient must be able to perform good oral hygiene
* With at least one implant with either cement or a screw-retained prosthesis demonstrating a diagnosis of peri-implantitis at an implant in function for a minimum of 1 year with a prosthesis installed.
* In cases where previous radiographic records are available: presence of bleeding and/or suppuration on gentle probing, increased probing depth compared to previous examinations, and radiographic evidence of bone loss beyond initial crestal remodeling. (Berglundh 2018).
* In cases where baseline radiographs are not available: presence of PPD ≥6 mm with BOP and/or suppuration (SUP) and radiographically detectable marginal bone loss (MBL) exceeding 3 mm on an implant in function forfor at least 1 year (Berglundh 2018).
* Target implants have to also demonstrate the presence of a peri-implant intra-bony defect with a depth ≥3 mm and width ≤4 mm, as assessed on radiographs and confirmed intra-surgically. In addition, the bony defect should present with a minimum of two walls .

No implant mobility and no evidence of occlusal overload. In patients presenting with more than one implant meeting the inclusion criteria, a single implant will be randomly selected for inclusion in the study.

Exclusion Criteria:

* Short implants (≤ 6mm)
* Contraindications for undergoing oral surgery.
* Patients pregnant or attempting to get pregnant (self-reported), or nursing women.
* Untreated/active periodontitis, or other untreated acute infections at the surgical site.
* Untreated malignancies at the surgical site.
* Self-reported current smoking, or active tobacco chewing, or chronic vaping.
* Taking long-term (>1yr) NSAID, prednisone or other anti-inflammatory prescription drugs
* Patients with any known history of blood disorders or complications such as abnormal concentration of thrombin and factor XIII in plasma, or hemophilia.
* Patients with significant co-morbidities, such as obesity, uncontrolled diabetes, immunosuppression, severe endocrine-induced bone diseases, signs of malnourishment, those receiving immunosuppressive therapy, poor tissue oxygenation or perfusion, and pre- or post-operative radiation.
* Unable to give consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic change | 12 months
  change in radiographic bone volume will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There are several patient level variables that can be used to identify the patient when used in combination.